CLINICAL TRIAL: NCT03458247
Title: Intra-individual Dose Escalation of Abiraterone Acetate According to Its Plasma Concentration in Patients With Progressive Castration-resistant Metastatic Prostate Cancer
Brief Title: Study of Dose Escalation of Abiraterone Actetate in Prostate Cancer
Acronym: OPTIMABI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Janssen, LP (Industry); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: P161201J; 2017-000560-15 (EudraCT Number)
Record Dates: First submitted 2018-02-02; First posted 2018-03-08 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Castration resistance; Drug monitoring; Abiraterone acetate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abiraterone acetate standard dose (Active Comparator): 1000 mg/day
  Interventions: Drug: Abiraterone acetate standard dose
- Abiraterone acetate escalated dose (Experimental): 2000 mg/day
  Interventions: Drug: Abiraterone acetate escalated dose

INTERVENTIONS:
Drug: Abiraterone acetate standard dose — 1000 mg/day
  Arms: Abiraterone acetate standard dose
Drug: Abiraterone acetate escalated dose — 2000 mg/day
  Arms: Abiraterone acetate escalated dose

SUMMARY:
The purpose of this study is to test whether a dose escalation up to 2000 mg per day of abiraterone acetate is feasible and lead to disease stabilization in castration-resistant metastatic prostate cancer patients who experience disease progression within the first 6 months of abiraterone actetate at standard dose (1000 mg/d) and have a plasma abiraterone concentration below 8.5 ng/mL.

It is a non-comparative phase 2 study in which patients will be included in two successive steps. Patients with mCRPC will be included in the first step and treated with standard dose (1000 mg/day) of ABI + prednisone /prednisolone (10 mg/d) according to the summary of product characteristics and monitored for trough ABI plasma level each month for 3 months.

In the second step intrapatient ABI dose escalation (2000 mg/day) + prednisone/prednisolone (10 mg/d) will be realized for patients from the first step experiencing progressive disease within 6 months of ABI standard dose and with mean ABI plasma level during the first three months < 8.5 ng/mL

DETAILED DESCRIPTION:
Metastatic castration-resistant prostate cancer (mCRPC) causes approximately 307,500 deaths annually worldwide. mCRPC has been defined as a clinical state in which, despite suppressed circulating testosterone levels lower than 50 ng/dL, the androgen receptor axis is reactivated. This reactivation is mainly due to the multiple signaling mechanisms in prostate cancer cells along with their microenvironment.

Thus, research efforts aimed at identifying new strategies to inhibit the androgen receptor axis. Abiraterone acetate (ABI) is a first-in-class inhibitor of cytochrome (CYP) 17A1, a critical enzyme for extra-gonadal and testicular androgen syntheses. ABI has shown impressive efficacy in treatment of mCRPC. ABI plus low-dose prednisone was first shown to improve survival in mCRPC patients pre-treated with docetaxel, and the combination therapy has since been approved for this purpose. Moreover, ABI plus low-dose prednisone resulted in prolonged overall survival (OS) as compared with placebo plus prednisone in docetaxel-naive patients. In these patients, ABI was associated with a median progression free survival of 16 months and median overall survival of 35 months. However, around 40% of patients do not experience PSA response to ABI therapy at 3 months. This parameter has been consistently identified as a surrogate parameter of time to progression.

As ABI is an oral agent that is subject to both inter- and intra-individual variability in bioavailability, its pharmacokinetics might be a critical parameter for its anticancer activity.

Investigators first established a simple method to mesure plasma ABI concentration by HPLC. They then conducted a prospective observational study in which they aimed to explore the relationship between ABI trough concentration and PSA response in mCRPC patients and to identify the critical determinants for its activity.

73 mCRPC patients, in whom treatment with ABI was indicated, were recruited from December 2012 to December 2014 in the oncology department of Cochin Hospital in Paris, France. The plasma concentration of ABI was determined at baseline, and then one (M1), two (M2) and three (M3) months after treatment initiation. The primary study objective was to investigate the relationship between ABI mean plasma trough concentration (ABI Cmin) and PSA response. PSA response was defined as a PSA decline of at least 50% after receiving ABI for 3 months.

In multivariate analysis, ABI Cmin was the only factor independently associated with PSA response: OR=1.12, [1.0-1.3], P=0.03. Based on these results, they established an optimal threshold of ABI C min by building a ROC curve. The treshold value of 8.45 ng/mL was associated with a specificity of and sensitivity of 70% [49-84] and 79% [63-81], respectively.

As plasma ABI exposure is a key element of PSA response, it supports the exploration of benefits of a pharmacokinetically-guided dosing strategy for ABI.

In a phase I trial, the recommended dose of ABI was 1000 mg per day as a plateau of endocrine effects was reported at doses greater than 750 mg. However, to their knowledge, no data regarding the effect of ABI on tissue androgens are available, and no dose limiting toxicity was identified up to 2000 mg per day which support the rational of a dose-escalation strategy. In a phase 2 study, 41 mCRPC patients received 1000 mg twice a day of ABI (2000 mg/day) and the tolerance profile appeared similar than with lower dose.

In this phase II trial, investigators aim to confirm the preliminary results presented above in a larger population. Moreover, their objective is to test whether a dose escalation up to 2000 mg per day is feasible and lead to disease stabilization in progressive patients within the first 6 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

Step 1

* Male 18 years and older.
* Voluntary signed informed consents of the patient before any study-specific procedure.
* Histologically confirmed prostate adenocarcinoma.
* Presence of bone and/or soft-tissue and/or visceral metastases through CT scan, MRI, scintigraphy scan.
* Progressive disease assessed by PSA, CT scan, MRI or bone scan according to the PCGW3 criteria PSA progression is defined as a 25% or greater increase and an absolute increase of 2 ng/mL or more from the nadir, which is confirmed by a second value obtained 1 or more weeks later. Bone scan: at least two or more new lesions are seen on bone scan compared with a prior scan.
* Patient with no or moderate symptoms (no need for continuous opioid treatment)
* Effective castration confirmed by testosterone plasma level < 50 ng/dL
* ECOG performance status: 0-2
* Life expectancy > 3 months
* Patient affiliate to french social assurance
* Laboratory criteria within 14 days before inclusion:

  * SGPT and SGOT < 5 fold the upper normal value
  * Kaliemia > 3 mM
* Patient using an effective contraceptive method during treatment

Step2

* Patients receiving ABI 1000 mg/day + prednisone/prednisolone 10 mg once a day through step 1 for at least two months
* At least two measures of ABI plasma concentrations available within the first three months of treatment
* Mean of ABI concentration < 8,5 ng/mL.
* Progressive disease occuring within 28 weeks following starting of ABI in the step 1. A progressive disease is assessed by PSA increase or bone scan according to PCWG3 criteria (15) or to CT scan according to RECIST 1.1 criteria (see § 2).
* Inclusion in step 2 must occur within 2 months following the first observation of cancer progression while in step 1.
* Patient using an effective contraceptive method during treatment

Exclusion Criteria:

Step 1

* Pure small cell carcinoma of the prostate or predominant histology of neuro-endocrine carcinoma.
* Confirmed brain and/or leptomeningeal metastases
* Previous treatment with docetaxel or any other anticancer treatment for castration-resistant prostate carcinoma (previous docetaxel for hormone-sensitive metastatic disease is allowed)
* Previous treatment with ABI or any other 17 B hydroxylase inhibitor or enzalutamide
* Treatment with first-generation antiandrogen (ciproterone acetate, bicalutamide, flutamide, nilutamide) performed on the day of baseline or within previous four weeks, due to possible anti-androgen withdrawal response. (This criterion does not apply for subjects, who have never responded to anti-androgen treatment).
* Patient co-morbidities:

  * Patients with the following hereditary diseases: galactose hypersensitivity, Lapp lactase deficiency.
  * Cirrhosis Child-Pugh B or C
  * Active or symptomatic viral hepatitis
  * Heart failure stage NYHA III or IV
  * Cardiac arythmia, heart failure stage NYHA II, ischemic cardiopathy or uncontroled hypertension, except if left ventricular ejection fraction is > 50%
  * Patients with left ventricular ejection fraction (LVEF) < 50%
  * Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment related complications.Prior or concurrent malignant disease in complete remission for less than 3 years, except T1N0 vocal cord carcinoma, basal or squamous cell skin carcinoma and in situ transitional cell bladder carcinoma
* Limitation of the patient's ability to comply with the treatment or to follow-up the protocol.

Step 2 Grade 3-4 toxicities related to ABI. In case of persistent grade 2 toxicity, inclusion in step 2 must be discussed in a case by case basis with the study coordinating Investigator.

* All non-inclusion criteria for step 1 applied
* Patient who is not adherent to ABI treatment at the investigator opinion
* Patient with a symptomatic and/or visceral tumor progression that would be an indication to start chemotherapy immediately according to the opinion of the investigator

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 94 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-12-27 (Actual)

PRIMARY OUTCOMES:
Non-progression rate | 12 weeks
  The proportion of patients who do not experience progressive disease (defined by PSA and/or radiographic progression) among those receiving ABI at a dose of 2000 mg / day + prednisone/prednisolone after failure of standard dose (1000 mg/day).

SECONDARY OUTCOMES:
Incidence of underexposure to ABI | 3 months
  Incidence of underexposure to ABI (mean plasma concentration < 8.5 ng/mL) in patients treated at standard dose (1000 mg / day) and identification of inter- and intra-individual variability factors of plasma levels of ABI
Evaluation of adherence to ABI and correlation with mean plasma ABI concentration | 3 months
  The adherence will be evaluated using two tools: the french version of the Girerd survey filled by the patient at 12 weeks and a personal treatment log book indicating daily times of drug administration
Evaluation of adherence to ABI and correlation with mean plasma ABI concentration | 6 months
  The adherence will be evaluated using two tools: the french version of the Girerd survey filled by the patient at 24 weeks and a personal treatment log book indicating daily times of drug administration
PSA response rate in patients treated at escalated dose | 6 months
  PSA response rate is defined as the proportion of patients with a decrease of ≥ 50% in the PSA concentration from the pretreatment baseline value, confirmed after ≥ 3 weeks by an additional PSA evaluation
Progression free survival in patients treated at escalated dose | 6 months
  Time from inclusion to progression or death in patients treated at escalated dose Disease progression is defined as either PSA or radiologic progression as described above
Incidence of adverse events related to ABI at a dose of 2000 mg/day according to the Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jerome ALEXANDRE, MD PhD, Study Director — Paris Descartes University, Assistance Publique Hôpitaux de Paris, Cochin hospital
Locations (1):
- Department of Medical Oncology, Cochin Hospital, Paris, paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexandre J, Oudard S, Golmard L, Campedel L, Mseddi M, Ladoire S, Khalil A, Maillet D, Tournigand C, Pasquiers B, Goirand F, Berthier J, Guitton J, Dariane C, Joly F, Xylinas E, Golmard JL, Abdoul H, Puszkiel A, Decleves X, Carton E, Thomas A, Vidal M, Huillard O, Blanchet B. Intra-individual Dose Escalation of Abiraterone According to Its Plasma Exposure in Patients with Progressive Metastatic Castration-Resistant Prostate Cancer: Results of the OPTIMABI Trial. Clin Pharmacokinet. 2024 Jul;63(7):1025-1036. doi: 10.1007/s40262-024-01396-x. Epub 2024 Jul 4. PMID 38963459
- [Background] Carton E, Noe G, Huillard O, Golmard L, Giroux J, Cessot A, Saidu NE, Peyromaure M, Zerbib M, Narjoz C, Guibourdenche J, Thomas A, Vidal M, Goldwasser F, Blanchet B, Alexandre J. Relation between plasma trough concentration of abiraterone and prostate-specific antigen response in metastatic castration-resistant prostate cancer patients. Eur J Cancer. 2017 Feb;72:54-61. doi: 10.1016/j.ejca.2016.11.027. Epub 2016 Dec 24. PMID 28027516